CLINICAL TRIAL: NCT00862641
Title: A Phase 4, Multi-Center, Double-Blind, Randomized, Placebo-Controlled Study of the Safety and Tolerance of Regadenoson in Subjects With Asthma or Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: A Study of the Safety and Tolerance of Regadenoson in Subjects With Asthma or Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 3606-CL-3001
Record Dates: First submitted 2009-03-15; First posted 2009-03-17 (Estimated); Results first posted 2010-12-15 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Asthma; Coronary Artery Disease; Pulmonary Disease, Chronic Obstructive
Keywords: regadenoson; CVT 3146; asthma; coronary artery disease; pulmonary disease, chronic obstructive
MeSH Terms: conditions — Asthma; Coronary Artery Disease; Pulmonary Disease, Chronic Obstructive | interventions — regadenoson

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo - Asthma (Placebo Comparator): Matching intravenous (IV) bolus injection, subjects with Asthma
  Interventions: Drug: Placebo
- Regadenoson - Asthma (Experimental): 0.4mg / 5mL intravenous bolus injection, subjects with Asthma
  Interventions: Drug: Regadenoson
- Placebo - COPD (Placebo Comparator): Matching intravenous bolus injection, subjects with Chronic Obstructive Pulmonary Disease (COPD)
  Interventions: Drug: Placebo
- Regadenoson - COPD (Experimental): 0.4mg / 5mL intravenous bolus injection, subjects with Chronic Obstructive Pulmonary Disease (COPD)
  Interventions: Drug: Regadenoson

INTERVENTIONS:
Drug: Regadenoson — IV
  Other Names: CVT3146; Lexiscan
  Arms: Regadenoson - Asthma; Regadenoson - COPD
Drug: Placebo — IV
  Arms: Placebo - Asthma; Placebo - COPD

SUMMARY:
This study is intended to determine the safety and tolerance of regadenoson in subjects with asthma or chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject has asthma or stable chronic obstructive pulmonary disease (COPD).
* Subject has a diagnosis of coronary artery disease (CAD) or risk factors for CAD as determined by a current medical diagnosis of at least 2 of the following conditions: Type 2 diabetes, hypertension, hypercholesterolemia, current or history of cigarette smoking (minimum 10 pack-years exposure) or obesity Body Mass Index (BMI > 30).
* Subject must abstain from smoking 3 hours prior and 8 hours post study drug administration.
* Subject must abstain from any intake of foods and beverages containing a methylated xanthine derivative (i.e. caffeine, theobromine, or methylxanthine) within 12 hours prior to study drug administration through the Follow-Up visit, as these foods may reduce the effects of regadenoson.
* Subject is able to safely abstain from theophylline for 12 hours prior to the Day 1 visit, as determined by the Investigator
* Asthma subject's frequency and severity of symptoms have remained unchanged within 30 days prior to study drug administration
* Asthma subject has FEV1 ≥60% predicted
* COPD subject has FEV1/FVC < 0.70

Exclusion Criteria:

* Female subject who is pregnant, lactating or of childbearing potential who refuses to use a medically acceptable form of contraception until the Follow-Up visit is complete.
* Subject started on a course of corticosteroids, steroid combination with long-acting Beta2-agonist (LABA) (oral or inhaled) or anticholinergic, or has undergone a change in dose of such medications ≤ 30 days prior to study drug administration (subject on a stable dose of such medications for > 30 days prior to study drug administration is allowed).
* Subject started leukotriene antagonists (e.g., montelukast), cromones (e.g., cromolyn sodium) or 5-lipoxygenase antagonists (e.g. zileuton or zyflo) or has undergone a change in dose of medications in these drug classes ≤ 7 days prior to study drug administration (subject on a stable dose of these medications for > 7 days prior to study drug administration is allowed).
* Subject has a history of second or third degree heart block or sinus node dysfunction unless the subject has a functioning pacemaker.
* Subject has symptomatic hypotension (temporary and reversible conditions that no longer exist are allowed).
* Subject is allergic or intolerant to aminophylline.
* Subject has had a respiratory infection within 2 weeks prior to randomization.
* Subject has had surgery within 3 months prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1009 (Actual)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Global Development
Locations (46):
- United States (46):
  - Montgomery, Alabama
  - Anaheim, California
  - Encinitas, California
  - Fullerton, California
  - Huntington Beach, California
  - Long Beach, California
  - Mission Viejo, California
  - Roseville, California
  - San Diego, California
  - Santa Ana, California
  - Waterbury, Connecticut
  - Newark, Delaware
  - Wilmington, Delaware
  - Clearwater, Florida
  - DeLand, Florida
  - Miami, Florida
  - Trinity, Florida
  - Winter Park, Florida
  - Stockbridge, Georgia
  - Aurora, Illinois
  - Topeka, Kansas
  - Shreveport, Louisiana
  - Auburn, Maine
  - No. Dartmouth, Massachusetts
  - Minneapolis, Minnesota
  - Plymouth, Minnesota
  - St Louis, Missouri
  - Papillion, Nebraska
  - Brick, New Jersey
  - Raleigh, North Carolina
  - Chardon, Ohio
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Upland, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Easley, South Carolina
  - Greenville, South Carolina
  - Spartanburg, South Carolina
  - Knoxville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - New Braunfels, Texas
  - San Antonio, Texas
  - Seattle, Washington

REFERENCES:
- [Result] Prenner BM, Bukofzer S, Behm S, Feaheny K, McNutt BE. A randomized, double-blind, placebo-controlled study assessing the safety and tolerability of regadenoson in subjects with asthma or chronic obstructive pulmonary disease. J Nucl Cardiol. 2012 Aug;19(4):681-92. doi: 10.1007/s12350-012-9547-4. Epub 2012 Apr 7. PMID 22484721
- See also: Link to Prescribing information — http://www.astellas.us/docs/lexiscan.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo - Asthma | Regadenoson - Asthma | Placebo - COPD | Regadenoson - COPD
Started | 177 | 360 | 152 | 320
Completed | 176 (Completed Population is equal to Safety Analysis Set (SAF)) | 356 (Completed Population is equal to Safety Analysis Set (SAF)) | 151 (Completed Population is equal to Safety Analysis Set (SAF)) | 316 (Completed Population is equal to Safety Analysis Set (SAF))
Not Completed | 1 | 4 | 1 | 4
Not completed — Randomized, but drug not received | 1 | 4 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo - Asthma | Regadenoson - Asthma | Placebo - COPD | Regadenoson - COPD | Total
Number analyzed (Participants) | 176 | 356 | 151 | 316 | 999
Age, Customized [Number; unit: participants]
  Between 18 and 64 years | 148 | 304 | 95 | 189 | 736
  >=65 years | 28 | 52 | 56 | 127 | 263
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 245 | 67 | 132 | 559
  Male | 61 | 111 | 84 | 184 | 440
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 128 | 283 | 136 | 284 | 831
  Black or African American | 45 | 61 | 13 | 22 | 141
  Asian | 1 | 4 | 0 | 6 | 11
  American Indian or Alaska Native | 1 | 6 | 2 | 1 | 10
  Native Hawaiian - Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Other | 1 | 2 | 0 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Had a >15% Decrease in Forced Expiratory Volume in 1 Second (FEV1) at the 2-hour Postbaseline Assessment
Description: FEV1 data was obtained by spirometry measures.
Time Frame: 2 Hours post dose
Population: The number of participants analyzed per arm represents Safety Analysis Set (SAF) which included all randomized subjects who received any amount of study drug.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Placebo - Asthma | Regadenoson - Asthma | Placebo - COPD | Regadenoson - COPD
Number analyzed (Participants) | 176 | 356 | 151 | 316
Percentage of Subjects | 2.9 | 1.1 | 5.4 | 4.2
Statistical Analysis 1: Comparison: Placebo - Asthma vs Regadenoson - Asthma; Test type: Superiority or Other; p = 0.1451, Cochran-Mantel-Haenszel; Analysis of treatment effect was based on the Cochran-Mantel Haenszel(CMH) test stratified by investigative site. Sites with <15 subjects were pooled
Statistical Analysis 2: Comparison: Placebo - COPD vs Regadenoson - COPD; Test type: Superiority or Other; p = 0.5790, Cochran-Mantel-Haenszel; Analysis of treatment effect was based on the CMH test stratified by investigative site. Sites with less than 15 subjects were pooled

2. Secondary Outcome: Use of Short-acting Bronchodilators for Treatment of Symptoms After Study Drug Administration
Description: The data represents the numbers of subjects using short acting bronchodilators at time of selected Adverse Event (AE).
  Short acting bronchodilators are defined as medications coded to drugs for obstructive airway disease.
  The selected respiratory symptomatic AEs included the following preferred terms: dyspnoea, dyspnoea exertional, obstructive airways disorder, tachypnoea, & wheezing.
Time Frame: Within 2 Hours of study drug administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Placebo - Asthma | Regadenoson - Asthma | Placebo - COPD | Regadenoson - COPD
Number analyzed (Participants) | 176 | 356 | 151 | 316
Subjects | 1 | 1 | 2 | 2

3. Secondary Outcome: Use of Short-acting Bronchodilators for Treatment of Symptoms After Study Drug Administration
Description: as for outcome 2
Time Frame: Within 24 Hours of study drug administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Placebo - Asthma | Regadenoson - Asthma | Placebo - COPD | Regadenoson - COPD
Number analyzed (Participants) | 176 | 356 | 151 | 316
Subjects | 2 | 5 | 2 | 5

4. Secondary Outcome: Change From Baseline to the 2 Hour Post-dose Assessment for FEV1 Absolute Values
Description: FEV1 data was obtained by spirometry measurements.
  Change from Baseline is calculated as the Hour 2 measurement minus the Baseline measurement.
Time Frame: Baseline and Hour 2
Population: The number of participants analyzed per arm represents Safety Analysis Set (SAF) which included all randomized subjects who received any amount of study drug. The number of participants included in the calculation for each time point is noted in the category titles, as "N".
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo - Asthma | Regadenoson - Asthma | Placebo - COPD | Regadenoson - COPD
Number analyzed (Participants) | 176 | 356 | 151 | 316
Liters
  Baseline (N=176; 356; 151; 316) | 2.41 (0.689) | 2.35 (0.623) | 1.70 (0.630) | 1.70 (0.655)
  Hour 2 (N=174; 351; 147; 313) | 2.37 (0.677) | 2.33 (0.615) | 1.69 (0.651) | 1.70 (0.647)
  Change at Hour 2 (N=174; 351; 147; 313) | -0.05 (0.160) | -0.01 (0.129) | -0.01 (0.152) | 0.00 (0.159)
Statistical Analysis 1: Comparison: Placebo - Asthma vs Regadenoson - Asthma; P-value applies to 'Change at Hour 2'; Test type: Superiority or Other; p = 0.0029, ANCOVA
Statistical Analysis 2: Comparison: Placebo - COPD vs Regadenoson - COPD; P-value applies to 'Change at Hour 2'; Test type: Superiority or Other; p = 0.6189, ANCOVA

5. Secondary Outcome: Change From Baseline to the 2 Hour Post-dose Assessment for FEV1 Percent Predicted
Description: as for outcome 4
Time Frame: Baseline and Hour 2
Population: The number of participants analyzed per arm represents Safety Analysis Set (SAF) which included all randomized subjects who received any amount of study drug. The number of participants included in the calculation for each row is noted in the category titles, as "N".
Measure: Mean (Standard Deviation); unit: Percentage of Predicted FEV1
Arm/Group | Placebo - Asthma | Regadenoson - Asthma | Placebo - COPD | Regadenoson - COPD
Number analyzed (Participants) | 176 | 356 | 151 | 316
Percentage of Predicted FEV1
  Baseline (N=176; 356; 151; 316) | 81.34 (13.679) | 80.32 (12.990) | 55.67 (15.131) | 55.69 (16.775)
  Hour 2 (N=174; 351; 147; 313) | 79.91 (13.591) | 80.11 (13.324) | 54.89 (15.601) | 55.61 (16.843)
  Change at Hour 2 (N=174; 351; 147; 313) | -1.56 (5.368) | -0.17 (4.519) | -0.56 (4.846) | -0.06 (5.170)
Statistical Analysis 1: Comparison: Placebo - Asthma vs Regadenoson - Asthma; P-value applies to 'Change at Hour 2'; Test type: Superiority or Other; p = 0.0015, ANCOVA
Statistical Analysis 2: Comparison: Placebo - COPD vs Regadenoson - COPD; P-value applies to 'Change at Hour 2'; Test type: Superiority or Other; p = 0.4385, ANCOVA

6. Secondary Outcome: Change From Baseline to the 2 Hour Post-dose Assessment for Forced Vital Capacity (FVC)
Description: FVC data was obtained by spirometry measurements.
  Change from Baseline is calculated as the Hour 2 measurement minus the Baseline measurement.
Time Frame: Baseline and Hour 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo - Asthma | Regadenoson - Asthma | Placebo - COPD | Regadenoson - COPD
Number analyzed (Participants) | 176 | 356 | 151 | 316
Liters
  Baseline (N=176; 356; 151; 316) | 3.22 (0.883) | 3.16 (0.829) | 2.75 (0.833) | 2.83 (0.889)
  Hour 2 (N=174; 351; 147; 313) | 3.17 (0.887) | 3.11 (0.809) | 2.70 (0.856) | 2.84 (0.857)
  Change at Hour 2 (N=174; 351; 147; 313) | -0.06 (0.208) | -0.03 (0.168) | -0.04 (0.230) | 0.00 (0.239)
Statistical Analysis 1: Comparison: Placebo - Asthma vs Regadenoson - Asthma; P-value applies to 'Change at Hour 2'; Test type: Superiority or Other; p = 0.0789, ANCOVA
Statistical Analysis 2: Comparison: Placebo - COPD vs Regadenoson - COPD; P-value applies to 'Change at Hour 2'; Test type: Superiority or Other; p = 0.0258, ANCOVA

7. Secondary Outcome: Change From Baseline to the 2 Hour Post-dose Assessment for FEV1/ FVC Ratio
Description: FEV1 and FVC data was obtained by spirometry measurements.
  Change from Baseline is calculated as the Hour 2 measurement minus the Baseline measurement.
Time Frame: Baseline and Hour 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of FEV1 / FVC
Arm/Group | Placebo - Asthma | Regadenoson - Asthma | Placebo - COPD | Regadenoson - COPD
Number analyzed (Participants) | 176 | 356 | 151 | 316
Percentage of FEV1 / FVC
  Baseline (N=176; 356; 151; 316) | 74.88 (7.510) | 74.59 (7.084) | 61.95 (12.684) | 60.00 (13.191)
  Hour 2 ( N=174; 351; 147; 313) | 75.11 (7.898) | 75.09 (7.074) | 62.26 (12.907) | 59.72 (13.171)
  Change at Hour 2 (N=174; 351; 147; 313) | 0.16 (3.329) | 0.52 (2.562) | 0.31 (3.177) | -0.30 (3.571)
Statistical Analysis 1: Comparison: Placebo - Asthma vs Regadenoson - Asthma; P-value applies to 'Change at Hour 2'; Test type: Superiority or Other; p = 0.2087, ANCOVA
Statistical Analysis 2: Comparison: Placebo - COPD vs Regadenoson - COPD; P-value applies to 'Change at Hour 2'; Test type: Superiority or Other; p = 0.0289, ANCOVA

8. Secondary Outcome: Change From Baseline to the 2 Hour Post-dose Assessment for Oxygen Saturation Measured by Pulse Oximetry
Description: Change from Baseline is calculated as the Hour 2 measurement minus the Baseline measurement.
Time Frame: Baseline and Hour 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of Oxygen Saturation
Arm/Group | Placebo - Asthma | Regadenoson - Asthma | Placebo - COPD | Regadenoson - COPD
Number analyzed (Participants) | 176 | 356 | 151 | 316
Percentage of Oxygen Saturation
  Baseline (N=170; 350; 143; 302) | 96.3 (1.81) | 96.3 (1.81) | 94.7 (2.40) | 95.0 (2.45)
  Hour 2 (N=170; 349; 143; 299) | 95.9 (1.80) | 96.0 (1.78) | 94.2 (2.25) | 94.5 (2.18)
  Change at Hour 2 (N=170; 349; 143; 299) | -0.4 (1.47) | -0.4 (1.35) | -0.4 (1.42) | -0.5 (1.66)
Statistical Analysis 1: Comparison: Placebo - Asthma vs Regadenoson - Asthma; P-value applies to 'Change at Hour 2' P-value based on ranked analysis of covariance with treatment and investigator site as main effects and baseline value as a covariate in the model; Test type: Superiority or Other; p = 0.9904, ANCOVA
Statistical Analysis 2: Comparison: Placebo - COPD vs Regadenoson - COPD; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.8085, ANCOVA

9. Secondary Outcome: Percentage of Selected Respiratory Adverse Events
Description: The selected respiratory Adverse Events are dyspnoea, dyspnoea exertional, obstructive airways disorder, tachypnoea and wheezing.
  Subjects may have reported more than one type of Adverse Event.
Time Frame: Within 24 Hours of study drug administration
Population: as for outcome 1
Measure: Number; unit: Percentage of Subjects
Arm/Group | Placebo - Asthma | Regadenoson - Asthma | Placebo - COPD | Regadenoson - COPD
Number analyzed (Participants) | 176 | 356 | 151 | 316
Percentage of Subjects
  Dyspnoea | 1.1 | 10.7 | 2.6 | 18.0
  Wheezing | 1.1 | 3.1 | 0.7 | 0.9
  Obstructive Airways Disorder | 0 | 0.3 | 0 | 0
  Dyspnoea Exertional | 0 | 0 | 0.7 | 0
  Tachypnoea | 0 | 0 | 0 | 0.3

ADVERSE EVENTS:
Time Frame: Adverse Event collection began immediately following study drug administration through the follow-up visit. Serious Adverse Events occurring until 30 days after dosing were reported.
Description: Treatment Emergent Adverse Events were defined as Adverse Events starting or worsening after starting administration of the test drug.
  Within a system organ class subjects may have reported more than one type of Adverse Event.
Arm/Group | Placebo - Asthma | Regadenoson - Asthma | Placebo - COPD | Regadenoson - COPD
Serious Adverse Events (participants affected / at risk) | 0/176 | 2/356 | 0/151 | 4/316
Other Adverse Events (participants affected / at risk) | 40/176 | 212/356 | 30/151 | 177/316
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Asthma (N=176) | Regadenoson - Asthma (N=356) | Placebo - COPD (N=151) | Regadenoson - COPD (N=316)
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Electrocardiogram change (Investigations) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — SAE was reported after the follow-up visit.
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 0 | 0 | 1 — SAE was reported after the follow-up visit.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Asthma (N=176) | Regadenoson - Asthma (N=356) | Placebo - COPD (N=151) | Regadenoson - COPD (N=316)
Headache (Nervous system disorders) | 17 | 97 | 12 | 62
Dizziness (Nervous system disorders) | 8 | 69 | 4 | 45
Dysgeusia (Nervous system disorders) | 13 | 33 | 6 | 29
Chest discomfort (General disorders) | 2 | 44 | 4 | 35
Feeling hot (General disorders) | 1 | 19 | 0 | 20
Tachycardia (Cardiac disorders) | 2 | 24 | 0 | 10
Palpitations (Cardiac disorders) | 0 | 19 | 1 | 11
Nausea (Gastrointestinal disorders) | 1 | 43 | 3 | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 38 | 4 | 57
Flushing (Vascular disorders) | 4 | 35 | 3 | 37
Heart rate increased (Investigations) | 0 | 20 | 0 | 15

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document. Sponsor may delay the publication for an additional 60 days to seek patent protection.